CLINICAL TRIAL: NCT06919627
Title: Negative HPV Test Results on Infinity/GeneXpert® With the Presence of a Late Amplification Signal: What Does This Mean ?
Brief Title: Negative HPV Test Results on Infinity/GeneXpert® With the Presence of a Late Amplification Signal: What Does This Mean ? (PaPCR)
Acronym: PaPCR
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC25.0053 - PaPCR
Record Dates: First submitted 2025-04-02; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-03

CONDITIONS: Cervical Cancers; Papillomavirus Infections; Papillomavirus Type 16/18 Infection
Keywords: papillomavirus; cancer; virology; PCR; GeneXpert; cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Papillomavirus Infections; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PCR HPV test with a late amplification signal in GeneXpert® : negative: Patients whose cervico-uterine sample was initially negative on the GeneXpert® system, but who had a late Ct signal (>35) on the initial gross result.
  Inclusion period: 01/01/2022 to 06/30/2024

SUMMARY:
The aim of this retrospective, single-center, observational study is to improve the diagnosis and interpretation of cervical cancer by better detection of epithelial lesions in the case of a late HPV PCR amplification signal rendered negative by routine laboratory testing using GeneXpert® technology.

The various evaluation criteria are :

* Presence or absence of lesions on cytological control following a negative HPV test with a late amplification signal on cervico-uterine and anal smear samples from patients seen in consultation at Brest University Hospital from 01/01/2022 to 30/06/2024 (after conventional PCR and genotyping).
* Comparison of the GeneXpert® technique with the results of another conventional pan-genotypic Papillomavirus PCR test.

DETAILED DESCRIPTION:
Cervical cancer is the fourth most common cancer in women worldwide, with 660,000 new cases and 350,000 related deaths by 2022. Papillomavirus (HPV) infection is the most common sexually transmitted infection in the world, and is transmitted by mucocutaneous contact. Incidence is particularly high in low- and middle-income countries, due to inadequate access to screening, treatment and vaccination against human papillomavirus (HPV). Numerous genotypes exist worldwide, some of which have oncogenic potential, principally genotypes 16, 18 and 45 (77% of all cervical cancers), and which should be screened as a priority by PCR.

In France, screening varies according to women's age: between the ages of 25 and 29, cytological examination is recommended every 3 years, following two initial tests carried out 1 year apart with normal results. Between the ages of 30 and 35, PCR detection of HPV at high risk of malignancy (HPV-HR) replaces cytological testing. This test is performed 3 years after the last normal cytological examination, and repeated every 5 years. If the PCR is positive, a cytological examination is performed. If the result is negative, a new PCR test is performed 1 year later.

The HPV test based on Cepheid® GeneXpert® technology detects HPV DNA, distinguishing between HPV 16 and 18/45, as well as other high-risk HPVs (31, 33, 35, 52, 58, 51, 59, 39, 56, 66, 68). The test targets E6/E7 oncogenes, and includes a sample adequacy check confirming the presence of human DNA in the sample. This quantitative real-time PCR test can provide quantitative information on viral load. A high viral load is a marker of persistent HPV infection, as well as a risk indicator for squamous intraepithelial lesions (SILs). However, the significance of low viral loads remains unclear.

GeneXpert® technology can produce "negative" results when late amplification (Ct approx. >37) is visible on qPCR curves.

It is difficult for medical biologists to biologically validate an uncertain result, so the aim of this study was to determine the significance of these late amplification curves using cytology results, as well as comparing GeneXpert® technology with in-house real-time PCR and genotyping in the event of positive samples.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose cervico-uterine swab was initially rendered negative by the GeneXpert® system when a late Ct signal (>35) was present in the raw result.

Exclusion Criteria:

* Patients with a positive cervico-uterine swab for Papillomavirus.
* Patients with a negative test with no amplification signal.
* Patients who have expressed opposition to inclusion in the study.
* Patients under legal protection (guardianship, curatorship, etc.).

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Women only (cervico-uterine sample tested)
Study Population: Patients who had a PCR HPV test with a late amplification signal in GeneXpert® and were found to be negative.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Age | 3 years
  in years
Date of sampling | 3 years
  DD/MM/YYYY
Cytology of sample | 3 years
  presence or absence of intraepithelial lesions
Clinical history | 10 years
  history of intraepithelial lesions or previous HPV test
Conization of lesions | 3 years
  yes or no
Treatment | 3 years
  yes or no

CONTACTS AND LOCATIONS:
Overall Officials: Christopher PAYAN, PU-PH, Principal Investigator — CHU de Brest
Locations (1):
- CHU de BREST, Brest, Brittany Region, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement